CLINICAL TRIAL: NCT04044339
Title: A Double-blind, Randomized, Placebo-controlled, Sponsor-open, Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TD-5202 in Healthy Subjects
Brief Title: Single and Multiple Ascending Dose, First-in- Human Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0177
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: TD-5202; 0177; single ascending dose; SAD; multiple ascending dose; MAD; first-in-human; Phase 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TD-5202 for SAD (Part A) (Experimental): 6 out of 8 subjects per cohort (up to 4 cohorts) will be randomized to receive TD-5202
  Interventions: Drug: TD-5202
- Placebo for SAD (Part A) (Placebo Comparator): 2 out of 8 subjects per cohort (up to 4 cohorts) will be randomized to receive placebo
  Interventions: Drug: Placebo
- TD-5202 for MAD (Part B) (Experimental): 6 out of 8 subjects per cohort (up to 3 cohorts) will be randomized to receive TD-5202
  Interventions: Drug: TD-5202
- Placebo for MAD (Part B) (Placebo Comparator): 2 out of 8 subjects per cohort (up to 3 cohorts) will be randomized to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-5202 — Study Drug to be administered orally
  Arms: TD-5202 for MAD (Part B); TD-5202 for SAD (Part A)
Drug: Placebo — Placebo to be administered orally
  Arms: Placebo for MAD (Part B); Placebo for SAD (Part A)

SUMMARY:
This is a Phase 1, randomized, double-blinded, placebo controlled study. The study consists of 2 parts: Part A is a single ascending dose (SAD) study in healthy subjects and Part B is a multiple ascending dose (MAD) study in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 19 - 55 years old
* Willing and able to give informed consent and comply with the study
* Medically healthy with no clinically significant medical history
* Body mass index (BMI) 18 to 32 kg/m2 and weighs at least 50 kg
* Women of child bearing potential must have a negative pregnancy test and use a highly efficient birth control method
* Males must use acceptable contraception
* Additional inclusion criteria apply

Exclusion Criteria:

* Positive for hepatitis A, B or C, HIV or tuberculosis
* Clinically significant abnormalities of laboratory evaluations
* Have abnormal ECG or vital sign measurements
* Any acute illness at time of screening
* Have a current bacterial, parasitic, fungal or viral infection
* Uses or have used tobacco or nicotine-containing products within 6 months prior to screening
* Additional inclusion criteria apply

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of SAD of TD-5202 by assessing the number, severity and type of treatment emergent adverse events | Day 1 through Day 8
To assess the safety and tolerability of MAD of TD-5202 by assessing the number, severity and type of treatment emergent adverse events | Day 1 through Day 17
Pharmacokinetics (PK) of TD-5202 when given as an SAD: AUC | Day 1 through Day 4
  Area under the plasma concentration-time curve (AUC)
Pharmacokinetics (PK) of TD-5202 when given as a SAD: Cmax | Day 1 through Day 4
  Maximum observed concentration (Cmax)
Pharmacokinetics (PK) of TD-5202 when given as a SAD: Tmax | Day 1 through Day 4
  Time to reach maximum observed concentration (Tmax)
PK of TD-5202 when given as an SAD: CL/F | Day 1 through Day 4
  Oral Clearance (CL/F)
PK of TD-5202 when given as an SAD: Vz/F | Day 1 through Day 4
  Terminal Phase Volume of Distribution(Vz/F)
PK of TD-5202 when given as an SAD: Kel | Day 1 through Day 4
  Elimination Rate (Kel)
PK of TD-5202 when given as an SAD: t 1/2 | Day 1 through Day 4
  Halflife (t 1/2)
PK of TD-5202 when given as an MAD: AUC | Day 1 and Day 10
  Area under the plasma concentration-time curve (AUC)
PK of TD-5202 when given as an MAD: Cmax | Day 1 and Day 10
  Maximum observed concentration (Cmax)
PK of TD-5202 when given as an MAD: Tmax | Day 1 and Day 10
  Time to reach maximum observed concentration (Tmax)
PK of TD-5202 when given as an MAD: C trough | Day 2, 4, 6, 8
  concentration at trough (after multiple dosing usually after reaching steady state) (C trough)
PK of TD-5202 when given as an MAD: Css | Day 10
  concentration at steady state (Css)
PK of TD-5202 when given as an MAD: CL/Fss | Day 10
  Oral clearance at steady state (CL/Fss)
PK of TD-5202 when given as an MAD: Cmin | Day 10
  Concentration minimum (after single dosing) (Cmin)
PK of TD-5202 when given as an MAD: Vz/Fss | Day 10
  Terminal phase volume of distribution at steady state (Vz/Fss)
PK of TD-5202 when given as an MAD: Kel | Day 10
  Elimination Rate (Kel)
PK of TD-5202 when given as an MAD: t 1/2 | Day 10
  Halflife (t 1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Theravance Biopharma Investigational Site, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.